CLINICAL TRIAL: NCT02829073
Title: Treating Tinnitus Using the Neuromonics Tinnitus Treatment Program: A Randomized, Double-blind Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Army Aeromedical Research Laboratory (U.S. Federal Agency)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, William A. Ahroon, Ph.D., Psychologist (Research), United States Army Aeromedical Research Laboratory
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USAARL 2014-045; IRB M-10464
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Tinnitus
Keywords: Tinnitus; Double-blind; Neuromonic Tinnitus Treatment Program; Oasis™
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oasis™ device (Experimental): Treatment using the Neuromonics Tinnitus Treatment Program and the Neuromonics Oasis™ treatment device.
  Interventions: Device: Neuromonics Tinnitus Treatment Program
- Placebo device (Placebo Comparator): Treatment using the Neuromonics Tinnitus Treatment Program and an identical-appearing placebo device.
  Interventions: Device: Placebo Device

INTERVENTIONS:
Device: Neuromonics Tinnitus Treatment Program — The Neuromonics Oasis™ treatment device will be fit to individuals reporting significant tinnitus. Assessment of primary and secondary measures will be made at 0 and 6 months following fitting.
  Other Names: Neuromonics Oasis™ treatment device
  Arms: Oasis™ device
Device: Placebo Device — A placebo device, identical to the Neuromonics Oasis™ device with altered firmware will be fit to individuals reporting significant tinnitus. Assessment of primary and secondary measures will be made at 0 and 6 months following fitting.
  Arms: Placebo device

SUMMARY:
The most current data indicate that tinnitus and hearing impairment are the Number 1 and 2 disabilities associated with service in Operations Iraqi Freedom and Enduring Freedom. Tinnitus can result from exposure to continuous noise from vehicles, generators, and other equipment, and from blast, or impulse noise from friendly-or opposing-forces weapon systems. Thus, tinnitus caused by both long-term noise exposure and acute acoustic trauma is an obstacle to be overcome in return-to-duty decisions and represents a serious liability to the retention of a healthy and fit force. Until recently, there has been no treatment that has been clinically validated as consistently effective. The development of the Neuromonics Tinnitus Treatment sought to overcome the practical limitations of previously available approaches (e.g. tinnitus maskers and biofeedback). While these studies have demonstrated the efficacy of the Neuromonics Tinnitus Treatment over alternative therapies, these trials studied target populations that may not be representative of the typical Soldier experiencing tinnitus.

One hundred and twenty (120) Soldiers or veterans with debilitating tinnitus will be recruited and divided into groups treated with two treatments, the Neuromonics Tinnitus Treatment Program which includes the use of the Neuromonics Oasis™ treatment device and a similarly-treated device using a placebo treatment. The study uses a randomized, double-blind design. The effectiveness of the treatments will be assessed using standard audiometric procedures and tinnitus subjective questionnaires.

This study will allow the Office of the Surgeon General of the Army to provide direction regarding the Neuromonics Tinnitus Treatment Program (NTTP) for alleviation of debilitating tinnitus that adversely affects Soldier deployability and operational performance. Retention of a fit force and improved quality of life for active-duty Soldiers are important issues associated with a successful approach to the treatment of tinnitus.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

Tinnitus, defined as the perception of sound when no corresponding external auditory stimulus exists, is a debilitating condition that is widespread yet difficult to successfully treat. It is estimated that between 10% and 15% of the adult population experience tinnitus to some degree. Although many people with tinnitus are not disturbed by the sensation, the condition is disabling in 0.5% to 2% of the tinnitus population or between 1.4 and 5 million people (Bauer & Brozoski, 2006). Additionally, tinnitus is among the most prevalent of service-connected disabilities for veterans receiving compensation according to the VA 2010 Annual Benefits Report, impacting over half a million veterans (US Department of Veterans Affairs, 2010).

The impact of tinnitus on a patient's quality of life can be devastating (Tyler & Baker, 1983). Many patients report that the intrusive perception of sound - such as ringing, roaring, or buzzing - interferes with their ability to relax, sleep and concentrate, especially in quiet situations. Many tinnitus patients also report reduced tolerance of loud sounds, and will tend to avoid noisy (e.g. social) situations. The disturbing effects of the condition can lead to a desperate sense of loss of control.

Until recently, there has been no treatment that has been clinically validated as consistently effective. Despite advances in understanding of the tinnitus condition, such as the Neurophysiological Model (Jastreboff & Hazell, 1993), the promise of much improved outcomes from treatment has yet to be realized in general clinical practice. Previously available treatment options continue to be limited by a lack of clinically consistent efficacy, efficiency, and/or user acceptability. Even Tinnitus Retraining Therapy (TRT), the most widely advocated practical application of the principles of the Neurophysiological Model, has been recently reported to yield only modest outcomes, and to require an extended period of time (up to 24 months) to achieve these outcomes for a high proportion of patients (J. A. Henry et al., 2005). Notably, some reports (Dineen, Doyle, Bench, & Perry, 1999; Hiller & Haerkotter, 2005; McKinney, Hazell, & Graham, 1999; Schmitt & Kroner-Herwig, 2002; Tyler, 2004) have questioned whether the acoustic stimulation used in tinnitus management programs such as TRT, predominantly consisting of broadband noise generators or hearing aids, provides any real incremental benefit over the counseling component of the program.

Furthermore, hearing aids and noise generators have been shown to provide limited clinical benefits when used in tinnitus management programs (Hiller & Haerkotter, 2005; Moffat et al., 2009), and these technologies are further limited by problems with user acceptability. Many tinnitus sufferers report that they find hearing aids intolerable to wear due to their decreased sound tolerance together with the unpredictability of amplified ambient sounds. Similarly, many people fitted with noise generators find the sound they produce unpleasant to listen to for the extended periods each day for which their use is recommended. As a result, for both hearing aids and noise generators, return-for-credit and "left-unused-in-the-drawer" rates are very high (J.A. Henry, Schecthter, Nagler, & Fausti, 2002; Hiller & Haerkotter, 2005).

Recent research into the pathogenesis of tinnitus has emphasized the role of neurological changes that result from damage to the auditory system (Tyler, 2005). These changes include the brain's adaptive response to auditory starvation (leading to increased sensitivity in the system), the initial perception of sound, and the systems within the brain that determine the person's attention and reaction to it.

The Neuromonics Tinnitus Treatment Program (NTTP) takes into account the neural plasticity that underlies tinnitus and targets the neurological changes that cause it. It utilizes an acoustic stimulus that combines music with an embedded neural stimulus, which are spectrally modified and customized for each patient's hearing and tinnitus profile. By accounting for a patient's hearing loss, the NTTP provides a broadband neural stimulus to stimulate the neural pathways that are "starved" due to auditory damage and/or hearing loss. The NTTP stimulus also positively engages the limbic system to reduce the stress caused by the tinnitus.

A key benefit of the customization process is that it allows the stimulus to be used at a comfortably low listening level. By allowing for intermittent, momentary perception of the tinnitus within a pleasant and relaxing listening experience, it desensitizes the patient's reaction to the tinnitus, thereby leading to long-term reduction in tinnitus disturbance.

The NTTP has been clinically proven in civilian populations to : (1) reduce symptoms early in treatment, in particular, provide relief from the disturbing effects of the condition, (2) treat the neurological causes associated with tinnitus, (3) provide long-term relief and improvements in quality of life, and (4) be convenient and noninvasive.

The NTTP has been the subject of a series of published clinical studies with civilian subjects (P. B. Davis, 2005; P. B. Davis, Paki, & Hanley, 2007; P.B. Davis, Wilde, & Steed, 2002; P. B. Davis, Wilde, Steed, & Hanley, 2008; Hanley, Davis, Paki, Quinn, & Bellekom, 2008), which have demonstrated that it yields better results, more quickly, more consistently, and with an intervention that is more acceptable to the patient than prior approaches. Included among these clinical studies was a comparative study (P. B. Davis et al., 2008) that showed that the Neuromonics Tinnitus Treatment generates significantly greater and more consistent improvements in tinnitus symptoms than a treatment comprised of counseling plus broad band noise ('white noise') and better outcomes than counseling-alone.

While the efficacy of the NTTP has been demonstrated, it remains an expensive and somewhat time-consuming treatment strategy. A previous study (Karch, Hill, Casto, Nedostup, & Staton, 2014) indicated that a COTS sound therapy may also be an effective way to treat tinnitus. Preliminary analysis of subjective tinnitus measures from Karch (2014) indicates that the NTTP strategies were effective at reducing the negative effects of tinnitus (i.e. reduction in subjective effects of tinnitus as measured by the Tinnitus Reaction Questionnaire (TRQ), tinnitus awareness time, and tinnitus disturbance time). Similar results were seen with a COTS group, with statistically significant differences in pre- and post-treatment measures of TRQ and tinnitus awareness. Analysis of clinical measures associated with tinnitus suggest no differences between pre- and post-treatment on the masking level required to cover tinnitus or the level of loudness discomfort associated with tinnitus for either group. However, due to the small sample size and unequal groups, comparisons between the treatments in the Karch et al. study (2014) should be made cautiously.

MILITARY RELEVANCE

Tinnitus is among the most prevalent medical complaints soldiers have when returning from Operation Iraqi Freedom/ Operation Enduring Freedom (OIF/OEF). Soldiers with clinically significant levels of tinnitus often suffer from anxiety, depression, sleep disruption, and difficulty concentrating. Currently, there is no standard tinnitus treatment protocol in the military system and limited clinical efficacy on the NTTP and COTS tinnitus treatment supported by a controlled study. The proposed research will attempt to definitively establish the value of the NTTP in a military setting.

The study stresses the return-to-duty of Soldiers experiencing severe tinnitus that might otherwise prevent these Soldiers from deploying with their units. Retention of a fit force and improved quality of life for active-duty Soldiers are important issues associated with a successful approach to the treatment of tinnitus.

OBJECTIVES/SPECIFIC AIMS/RESEARCH QUESTIONS

The objective of the study is to determine the effectiveness of individualized sound stimuli used in a FDA classified tinnitus masker device, the Neuromonics, Inc. Oasis™.

Research Question: Is there a difference in clinical outcomes for tinnitus patients treated with the NTTP compared with the same treatment using a placebo-control device? The placebo-control device is otherwise identical to the NTTP device except that the sound stimuli are not matched to the patients' audiograms and tinnitus profile and are not specifically designed to promote relaxation. Assignment of tinnitus patients to the treatment and placebo groups is performed off site and the experimenters have no information on group assignment.

Hypothesis: In the Active Duty, Reserve, and National Guard military and recently separated veteran populations with complaints of tinnitus, the NTTP group will have significantly improved tinnitus clinical outcomes in comparison to placebo-control group at 6 months. Clinical outcomes are described in Section B5.4 and Table 1 below.

Null Hypothesis: In the Active Duty, Reserve, and National Guard military and recently separated veteran populations with complaints of tinnitus, the NTTP group will have tinnitus clinical outcomes statistically indistinguishable from the placebo-control group at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* If an active duty military personnel, must be between the ages of 18 to 60 years at the time of enrollment.
* If a veteran, must be between the ages of 19 to 60 years at the time of enrollment
* Tinnitus disturbance determined at the initial pre-enrollment assessment to be clinically significant, as denoted by a score on the TRQ of 17-70; and
* Four frequency (0.5, 1, 2, and 4 kHz) pure tone average in one ear (0.5, 1, 2, and 4 kHz) is equal to or less than 50dB HL, as determined by audiometry performed at the initial pre-enrollment assessment; and
* Cognitive, comprehension and manual dexterity abilities sufficient to self-administer treatment, and ability to travel to attend appointments, as necessary, as determined at the initial pre-enrollment assessment; and
* Motivated to pursue treatment and has appropriate expectations as to treatment outcomes (including the possibility of being assigned to the placebo group), as determined at the initial pre-enrollment assessment.
* Must have access to healthcare for follow-up care for the six month study period

Exclusion Criteria:

* Refusal to give consent
* Significant psychological disturbance [defined as any rating other than 0 on Question Number 24 the TRQ (suicidal ideology) or a score of more than 78 on the Tinnitus Handicap Inventory (THI)] that may interfere with the treatment as assessed by the treating clinician and/or referring physician;
* Complicating medical conditions such as acute/unstable Meniere's disease as inferred by responses on the Tinnitus History Questionnaire (THQ);
* Ongoing use of ototoxic medications (THQ);
* Pulsatile tinnitus (THQ);
* Continued excessive noise exposure without effective hearing protection (THQ);
* After all elements of informed consent are completed and the TRQ has been scored, a score of less than 17 will exclude the volunteer from participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Reaction Questionnaire (TRQ) | Baseline and two, four, and six months after enrollment
  Change in TRQ score at 6 months compared to baseline

SECONDARY OUTCOMES:
Tinnitus Reaction Questionnaire (TRQ) Midterm | Baseline and two, four, and six months after enrollment
  Change in TRQ score at 2 and 4 months compared to baseline
Tinnitus Reaction Questionnaire (TRQ) Awareness | Baseline and two, four, and six months after enrollment
  Change of tinnitus awareness at 2, 4, and 6 months compared to baseline
Tinnitus Reaction Questionnaire (TRQ) Bothersome | Initial and two, four, and six months after enrollment
  Change of bothersome tinnitus at 2, 4, and 6 months compared to baseline
PTSD Checklist-Military (PCL-M) | Baseline and two, four, and six months after enrollment
  Change in PLC-M score at 2, 4, and 6 months compared to baseline
Hospital Anxiety and Depression Scale (HADS) | Baseline and six months after enrollment
  Change in HADS score at 6 months compared to baseline
Minimum Masking Level (MML) (an audiometric test) | Baseline and six months after enrollment
  Change in MML at 6 months compared to baseline
Loudness Discomfort Levels (LDL) (an audiometric test) | Baseline and six months after enrollment
  Change in LDL at 6 months compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: William A Ahroon, Ph.D., Principal Investigator — U.S. Army Aeromedical Research Laboratory
Locations (1):
- U.S. Army Aeromedical Research Laboratory, Fort Rucker, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis PB, Paki B, Hanley PJ. Neuromonics Tinnitus Treatment: third clinical trial. Ear Hear. 2007 Apr;28(2):242-59. doi: 10.1097/AUD.0b013e3180312619. PMID 17496674
- [Background] Davis PB, Wilde RA, Steed LG, Hanley PJ. Treatment of tinnitus with a customized acoustic neural stimulus: a controlled clinical study. Ear Nose Throat J. 2008 Jun;87(6):330-9. PMID 18561116
- [Background] Hanley PJ, Davis PB, Paki B, Quinn SA, Bellekom SR. Treatment of tinnitus with a customized, dynamic acoustic neural stimulus: clinical outcomes in general private practice. Ann Otol Rhinol Laryngol. 2008 Nov;117(11):791-9. doi: 10.1177/000348940811701101. PMID 19102123
- [Background] Karch, S.J., et al., Evaluation of Sound Therapy Tinnitus Treatments with Concurrent Counseling in Active Duty Military Personnel. 2014, U.S. Army Aeromedical Research Laboratory: Fort Rucker, AL.
- [Background] Bauer CA, Brozoski TJ. Effect of gabapentin on the sensation and impact of tinnitus. Laryngoscope. 2006 May;116(5):675-81. doi: 10.1097/01.MLG.0000216812.65206.CD. PMID 16652071
- [Background] Tyler RS, Baker LJ. Difficulties experienced by tinnitus sufferers. J Speech Hear Disord. 1983 May;48(2):150-4. doi: 10.1044/jshd.4802.150. PMID 6621006
- [Background] Jastreboff PJ, Hazell JW. A neurophysiological approach to tinnitus: clinical implications. Br J Audiol. 1993 Feb;27(1):7-17. doi: 10.3109/03005369309077884. PMID 8339063
- [Background] Henry JA, Schechter MA, Loovis CL, Zaugg TL, Kaelin C, Montero M. Clinical management of tinnitus using a "progressive intervention" approach. J Rehabil Res Dev. 2005 Jul-Aug;42(4 Suppl 2):95-116. doi: 10.1682/jrrd.2005.01.0005. PMID 16470467
- [Background] Dineen R, Doyle J, Bench J, Perry A. The influence of training on tinnitus perception: an evaluation 12 months after tinnitus management training. Br J Audiol. 1999 Feb;33(1):29-51. doi: 10.3109/03005364000000098. PMID 10219721
- [Background] Hiller W, Haerkotter C. Does sound stimulation have additive effects on cognitive-behavioral treatment of chronic tinnitus? Behav Res Ther. 2005 May;43(5):595-612. doi: 10.1016/j.brat.2004.03.012. PMID 15865915
- [Background] Moffat G, Adjout K, Gallego S, Thai-Van H, Collet L, Norena AJ. Effects of hearing aid fitting on the perceptual characteristics of tinnitus. Hear Res. 2009 Aug;254(1-2):82-91. doi: 10.1016/j.heares.2009.04.016. Epub 2009 May 3. PMID 19409969
- [Background] Karch, S. J., Hill, M. M., Casto, K. L., Nedostup, A. E., & Staton, R. N. (2014). Evaluation of Sound Therapy Tinnitus Treatments with Concurrent Counseling in Active Duty Military Personnel. (Report 2014-022). Fort Rucker, AL: U.S. Army Aeromedical Research Laboratory.
- [Background] US Department of Veterans Affairs. (2010). 2010 Annual Benefits Report. Retrieved from www.vba.va.gov/REPORTS/abr/2010_abr.pdf.
- [Background] McKinney, C.J., J.W. Hazell, and R.L. Graham, An evaluation of the TRT method, in Proceedings of the sixth international tinnitus seminar, J.W. Hazell, Editor. 1999. p. 99-105.
- [Background] Schmitt, C. and B. Kroner-Herwig, Comparison of tinnitus coping training and TRT: Are they superior to education?, in Proceedings of the Seventh International Tinnitus Seminar, R. Patuzzi, Editor. 2002, Hawthorn Production Services: Norfolk, VA. p. 273-276.
- [Background] Tyler, R.S., Final Report: A preliminary investigation of the effectiveness of tinnitus retraining therapy. Tinnitus Today, 2004. 29: p. 12.
- [Background] Henry, J.A., et al., Tinnitus retraining therapy and masking; how do they compare?, in Proceedings of the Seventh International Tinnitus Seminar, R. Patuzzi, Editor. 2002, Hawthorn Production Services: Norfolk, VA. p. 247-254.
- [Background] Tyler, R.S., Neurophysiological models, psychological models, and treatments for tinnitus, in Tinnitus Treatments: Clinical Protocols, R.S. Tyler, Editor. 2005, Thieme Medical Publishers: New York. p. 1-22.
- [Background] Davis, P.B., R.A. Wilde, and L.G. Steed. Clinical trial findings of a neurophysiologically-based tinnitus rehabilitation technique using tinnitus desensitization music. in Proceedings of the Seventh International Tinnitus Seminar. 2002. Perth: University of Western Australia.
- [Background] Davis, P.B., Music and the acoustic desensitization protocol for tinnitus., in Tinnitus treatments R.S. Tyler, Editor. 2005, Thieme: New York.